CLINICAL TRIAL: NCT03977298
Title: Surgical Protocol for Peri-implantitis in Vertical Defect in Absence of Keratinised Tissue Using Chemical Decontamination With Chlorexidine and a CTG: a Randomized Clinical Trial
Brief Title: Surgical Protocol for Peri-Implantitis Treatment-4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Clementini, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: peri-implant surgical-4
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; CTG; Chlorhexidine; surgical treatment; Keratinised tissue
MeSH Terms: conditions — Peri-Implantitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Sham Comparator): Access flap will be raised to gain access to the implant surface. Inflammatory tissue, excess cement or plaque deposits will be removed using titanium curettes and the implant surface will be cleaned by copious irrigation with sterile saline and surgical gauze soaked in Chlorhexidine
  Interventions: Procedure: Chlorhexidine
- Connective Tissue Graft (Other): CTG will be positioned in the buccal aspect of the peri-implant tissue
  Interventions: Procedure: Chlorhexidine; Procedure: CTG

INTERVENTIONS:
Procedure: Chlorhexidine — Inflammatory tissue, excess cement or plaque deposits will be removed using titanium curettes and the implant surface will be cleaned by copious irrigation with sterile saline and surgical gauze soaked in chlorhexidine
Procedure: CTG — CTG will be positioned in the buccal aspect of the peri-implant tissue
  Arms: Connective Tissue Graft

SUMMARY:
Peri-implant diseases are common post-restorative complications in implant rehabilitations and they occur with an incidence of 12-43%.

Based on the available data in literature, the surgical therapy for peri-implantitis is effective in disease resolution. Surgical access to peri-implant lesions facilitates the removal of all granulation tissue from the defect area as well as debridement and decontamination of the exposed implant surface defect area.

Different techniques have been used for implant surface decontamination during peri-implant surgery, including mechanical, chemical and laser treatments.

DETAILED DESCRIPTION:
Peri-implantitis are defined as inflammatory diseases caused by bacterial biofilm around implant surface characterized by bleeding on probing, probing depth and eventually bone loss; if not successfully treated they may lead to implant loss. Based on the available parameters that have been reported in literature non surgical therapy doesn't seem to be effective on peri-implantitis.

Therefore it is recommended to consider advanced therapies such as surgical interventions when non surgical peri-implant therapy fails to achieve significant improvements in clinical parameters. Numerous approaches have been used for implant surface decontamination during per-implant surgery, including mechanical, chemical and laser treatments. Conventional mechanical means don't seem to be effective on peri-implant diseases. In addition, the rough implant surface is a retentive factor for bacterial colonization and therefore makes implant surface difficult to debride. Another problem in maintaining implant health concerns the presence or absence of keratinised tissue around implant: if present, it seams to help the patient to maintain an optimal level of oral hygiene around implant and therefore the implant survival itself.

The aim of the present randomized controlled clinical trial is to assess the influence of keratinised tissue around implant in improving clinical parameters. In particular, implant surface will be decontaminated mechanically with titanium curettes and chemically using chlorhexidine; after this the bone defect will be filled with bio-materlal and a CTG around tissue implant will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one screw-type titanium implant exhibiting bleeding and/or suppuration on probing combined with:

  1. PPD ≥ 5 mm and bone loss ≥ 2 mm (compared to crestal bone levels at the time of placement of the reconstruction)
  2. PPD ≥6 and bone loss ≥3 (not compared to crestal bone levels at the time of placement of the reconstruction)
* single tooth and bridgework restorations without overhangs no evidence of occlusal overload (i.e. occlusal contacts revealed appropriate adjustment)
* treated chronic periodontitis and proper periodontal maintenance care FMPS < 20%
* non-smoker or light smoking status in smokers (<10 cigarettes per day) implant function time ≥ 1 year.

Exclusion Criteria:

* Patients with uncontrolled diabetes
* patients with osteoporosis or under bisphosphonate medication,
* pregnant or lactating women
* patients with a history of radiotherapy to the head and neck region hollow implants
* implant mobility
* implants at which no position could be identified where proper probing measurements could be performed;
* previous surgical treatment of the peri-implantitis lesions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing changes | baseline, 3, 6 and 12 months after treatment
  changes of bleeding on probing, evaluated as present if bleeding will be evident within 30 s after probing, or absent, if no bleeding will be noticed within 30 s after probing

SECONDARY OUTCOMES:
clinical attachment level changes | baseline, 3, 6 and 12 months after treatment
  changes in clinical attachment level, measured from CEJ to the tip of the probe
probing pocket depth changes | baseline, 3, 6 and 12 months after treatment
  changes in probing depth probing, measured from gingival margin to te tip of the probe
mucosal recession changes | baseline, 3, 6 and 12 months after treatment
  changes in mucosal recession, measured from CEJ to gingival margin
bone level changes | baseline, 3, 6 and 12 months after treatment
  changes in bone level at mesial and distal aspect, measured on periapical X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, Study Chair — Università Vita-Salute San Raffaele
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Italy